CLINICAL TRIAL: NCT02215252
Title: A Randomized Double Blind Placebo And Active Controlled Parallel Group Phase 2 Study To Evaluate PF-05089771 As A Monotherapy And As An Add-on To Pregabalin For The Treatment Of Painful Diabetic Peripheral Neuropathy
Brief Title: A Clinical Trial To Evaluate PF-05089771 On Its Own And As An Add-On Therapy To Pregabalin (Lyrica) For The Treatment Of Pain Due To Diabetic Peripheral Neuropathy (DPN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3291026; DPN NAV1.7 (Other: Alias Study Number)
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — PF-05089771; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PF-05089771 (Experimental)
  Interventions: Drug: PF-05089771 150 mg
- Placebo (Experimental)
  Interventions: Drug: Matched placebo for PF-05089771 150 mg and pregabalin 300 mg
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin 300 mg
- PF-05089771 + Pregabalin (Experimental)
  Interventions: Drug: PF-05089771 150 mg + Pregabalin 300 mg

INTERVENTIONS:
Drug: PF-05089771 150 mg — PF-05089771 150 mg twice daily oral dosing with capsules. Treatment period = 4 weeks.
  Arms: PF-05089771
Drug: Matched placebo for PF-05089771 150 mg and pregabalin 300 mg — Matched placebo for PF-05089771 150 mg twice daily and pregabalin 150 mg twice daily oral dosing with capsules. Treatment period = 4 weeks.
  Arms: Placebo
Drug: Pregabalin 300 mg — Pregabalin 150 mg twice daily oral dosing with capsules. Treatment period = 4 weeks.
  Arms: Pregabalin
Drug: PF-05089771 150 mg + Pregabalin 300 mg — PF-05089771 150 mg twice daily oral capsules with pregabalin 150 mg twice daily oral capsules. Treatment period = 4 weeks.
  Arms: PF-05089771 + Pregabalin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PF-05089771 as a monotherapy and as an add-on to pregabalin for the treatment of painful diabetic peripheral neuropathy (DPN)

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years to 80 years.
* Diagnosis of Type 2 diabetes mellitlus (T2DM) with current glycosylated hemoglobin A1c (HbA1c) levels of ≤ 11% at Screening and on a stable antidiabetic medication regimen for at least 30 days prior to randomization.
* Presence of ongoing pain due to DPN for at least 6 months.
* Willing to discontinue protocol-specified prohibited pain medications for DPN throughout the duration of the study.

Exclusion Criteria:

* Painful neuropathies or painful conditions other than DPN that may confound evaluation of pain due to DPN during the study.
* Subjects who have failed previously on pregabalin (at the recommended label dose and for adequate duration) due to lack of efficacy.
* Subjects with any clinically significant medical or psychiatric conditions or clinically significant laboratory test abnormalities.
* Pregnant women, lactating mothers, men with partners currently pregnant, women suspected of being pregnant, and women who wish to be pregnant during the course of the clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2014-11-10 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (32):
  - Clinical Research Consortium Arizona, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Neuro-Pain Medical Center, Fresno, California
  - Meridien Research, Bradenton, Florida
  - PAB Clinical Research, Brandon, Florida
  - Pulmonary Associates of Brandon (PAB), Brandon, Florida
  - Meridien Research, Brooksville, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - MD Clinical, Hallandale, Florida
  - Meridien Research, Lakeland, Florida
  - Family Care Specialists, Ocala, Florida
  - Renstar Medical Research, Ocala, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Metabolic Research Institute, Inc, West Palm Beach, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Clinical Research Advantage, Inc, Evansville, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Novex Clinical Research, LLC, New Bedford, Massachusetts
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Consortium, Las Vegas, Nevada
  - The Medical Research Network, LLC, New York, New York
  - New Phase Research and Development, Knoxville, Tennessee
  - Internal Medicine Associates, Tullahoma, Tennessee
  - Trinity Clinical Research, LLC, Tullahoma, Tennessee
  - KRK Medical Research, Arlington, Texas
  - Nerve and Muscle Center of Texas, Houston, Texas
  - National Clinical Research - Norfolk, Inc, Norfolk, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Rainier Clinical Research Center, Inc, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3291026&StudyName=A%20Clinical%20Trial%20To%20Evaluate%20PF-05089771%20On%20Its%20Own%20And%20As%20An%20Add-On%20Therapy%20To%20Pregabalin%20%28Lyrica%29%20For%20The%20Treatment%20Of%20Pain%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility included healthy male and/or female participants of non childbearing potential between the ages of 18 and 80 years, inclusive, and a diagnosis of painful diabetic peripheral neuropathy and type II diabetes.
  Following the interim analysis, the study was stopped. No participants were dosed with PF-05089771 150mg BID + pregabalin.
Pre-assignment Details: A number of 141 participants were the anticipated to be enrolled based on a discontinuation rate calculated from previous Pfizer DPN studies.
  The study discontinuation rate was lower than anticipated, hence fewer participants were randomized.
Groups:
- PF-05089771 150 mg BID: Participants received PF-05089771 150mg oral capsules twice daily (BID) for 4 weeks.
- Pregabalin: Participants received pregabalin, oral capsule, 150 mg/day, then 300 mg/day from Day 8, for 4 weeks.
- Placebo: Participants received matched placebo oral capsule for 4 weeks.
Period: Overall Study
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Started | 44 | 46 | 45
Completed | 42 | 38 | 41
Not Completed | 2 | 8 | 4
Not completed — Adverse Event | 1 | 5 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Does not Meet Entrance Criteria | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Other | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo | Total
Number analyzed (Participants) | 44 | 46 | 45 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.4) | 58.1 (11.3) | 59.2 (10.9) | 58.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 14 | 50
  Male | 27 | 27 | 31 | 85

OUTCOME MEASURES:

1. Primary Outcome: Daily Pain Numeric Rating Scale (NRS)
Description: The endpoint average pain score, based on the mean of the last 7 days' daily pain numeric rating scale (NRS) scores at (NRS is an 11-point scale where 0 = no pain and 10 = worst possible pain) from the daily pain diaries while receiving study medication during the treatment period.
Time Frame: Baseline, Week 1, Week 2, Week 3 and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Unit on a scale
  Baseline (n = 44, 46, 45) | 6.17 (1.164) | 6.62 (1.420) | 6.35 (1.170)
  Week 1 (n = 44, 46, 44) | 5.45 (1.372) | 5.87 (1.872) | 6.07 (1.454)
  Week 2 (n = 43, 44, 40) | 5.14 (1.762) | 5.26 (2.302) | 6.10 (1.504)
  Week 3 (n = 38, 40, 41) | 5.01 (1.820) | 5.36 (2.386) | 5.76 (1.540)
  Week 4 (n = 41, 38, 39) | 4.83 (1.595) | 5.14 (2.508) | 5.61 (1.820)
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for week 4. Mixed Models Repeated Measures analysis including all data up to Week 4 ,incorporating Bayesian priors separately on the placebo response and pregabalin effect; Test type: Superiority or Other; Mean Difference (Final Values) = -0.41, 90% CI 2-sided [-1.00 to 0.17], Standard Deviation 0.355
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.53, 90% CI 2-sided [-0.91 to -0.20], Standard Deviation 0.230

2. Secondary Outcome: Responder Rate Based on a 30% Improvement in Mean Pain Response Using the Daily Pain NRS Score
Description: Percentage of participants that received ≥30% improvement from baseline in mean pain response (from the daily pain diary).
Time Frame: Baseline, Week 1, Week 2, Week 3 and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Percentage of participants
  Week 1 (n = 44, 46, 45) | 9.09 | 15.22 | 4.44
  Week 2 (n = 44, 45, 44) | 22.73 | 31.11 | 9.09
  Week 3 (n = 42, 42, 43) | 23.81 | 26.19 | 11.63
  Week 4 (n = 42, 38, 43) | 28.57 | 31.58 | 16.28
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Logistic Regression using all data up to Week 4; Test type: Superiority or Other; Odds Ratio (OR) = 1.91, 90% CI 2-sided [0.78 to 4.69]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Logistic Regression using all data up to Week 4; Test type: Superiority or Other; Odds Ratio (OR) = 2.63, 90% CI 2-sided [1.06 to 6.56]

3. Secondary Outcome: Responder Rate Based on a 50% Improvement in Mean Pain Response Using the Daily Pain NRS Score
Description: Percentage of participants that received ≥50% improvement from baseline in mean pain response (from the daily pain diary).
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Percentage of participants
  Week 1 (n = 44, 46, 45) | 0 | 4.35 | 4.44
  Week 2 (n = 44, 45, 44) | 11.36 | 15.56 | 2.27
  Week 3 (n = 42, 42, 43) | 7.14 | 19.05 | 2.33
  Week 4 (n = 42, 38, 43) | 9.52 | 23.68 | 6.98
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Logistic Regression using all data up to Week 4; Test type: Superiority or Other; Odds Ratio (OR) = 1.25, 90% CI 2-sided [0.33 to 4.74]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Logistic Regression using all data up to Week 4; Test type: Superiority or Other; Odds Ratio (OR) = 4.75, 90% CI 2-sided [1.43 to 15.81]

4. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) - Burning (Superficial) Spontaneous Pain
Description: Participants rated questionnaire to evaluate different symptoms of neuropathic pain (dimensions: burning [superficial] spontaneous pain, pressing [deep] spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dyesthesia [P/D]) including 10 descriptors quantified on a 0 (no symptoms) to 10 (worst symptoms imaginable) and 2 temporal items assessing duration of spontaneous ongoing and paroxysmal pain. A score in each dimension and also a total score (from 0-100) is generated using data from the questionnaire. Higher score indicates a greater intensity of pain.
Time Frame: Baseline, Week 2, and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Unit on a scale
  Baseline (n = 44, 46, 45) | 4.6 (2.71) | 5.3 (2.49) | 4.8 (2.35)
  Week 2 (n = 42, 41, 43) | 3.7 (2.94) | 4.3 (3.06) | 4.2 (2.35)
  Week 4 (n = 42, 38, 42) | 3.4 (3.04) | 4.3 (2.80) | 4.5 (2.55)
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -1.04, 90% CI 2-sided [-1.75 to -0.32], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -0.69, 90% CI 2-sided [-1.43 to 0.04], Standard Error of Mean 0.44

5. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) - Pressing (Deep) Spontaneous Pain
Description: Participant rated questionnaire to evaluate different symptoms of neuropathic pain (dimensions: burning [superficial] spontaneous pain, pressing [deep] spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dyesthesia [P/D]) including 10 descriptors quantified on a 0 (no symptoms) to 10 (worst symptoms imaginable) and 2 temporal items assessing duration of spontaneous ongoing and paroxysmal pain. A score in each dimension and also a total score (from 0-100) is generated using data from the questionnaire. Higher score indicates a greater intensity of pain.
Time Frame: Baseline, Week 2 and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Unit on a scale
  Baseline (n = 44, 46, 45) | 3.8 (2.48) | 4.9 (2.21) | 4.5 (2.40)
  Week 2 (n = 42, 41, 43) | 3.3 (2.51) | 4.4 (2.83) | 4.2 (2.33)
  Week 4 (n = 42, 38, 42) | 3.4 (2.67) | 3.9 (3.08) | 4.0 (2.48)
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -0.22, 90% CI 2-sided [-0.86 to 0.43], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -0.66, 90% CI 2-sided [-1.33 to 0.00], Standard Error of Mean 0.40

6. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) - Paroxysmal Pain
Description: as for outcome 5
Time Frame: Baseline, Week 2, and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Unit on a scale
  Baseline (n = 44, 46, 45) | 4.5 (2.36) | 5.8 (2.18) | 5.6 (2.23)
  Week 2 (n = 42, 41, 43) | 4.1 (2.61) | 4.7 (2.98) | 4.9 (2.11)
  Week 4 (n = 42, 38, 42） | 3.9 (2.87) | 4.6 (2.83) | 4.8 (2.55)
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -0.10, 90% CI 2-sided [-0.87 to 0.67], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -0.58, 90% CI 2-sided [-1.36 to 0.20], Standard Error of Mean 0.47

7. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) - Evoked Pain
Description: as for outcome 5
Time Frame: Baseline, Week 2 and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Unit on a scale
  Baseline (n = 44, 45, 45) | 2.7 (2.38) | 5.0 (2.51) | 4.2 (2.42)
  Week 2 (n = 42, 40, 43) | 2.0 (1.92) | 4.0 (2.67) | 3.5 (2.47)
  Week 4 (n = 42, 37, 42) | 2.3 (2.24) | 3.8 (3.07) | 3.6 (2.53)
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = 0.09, 90% CI 2-sided [-0.49 to 0.67], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -0.46, 90% CI 2-sided [-1.05 to 0.13], Standard Error of Mean 0.36

8. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) - Paresthesia/Dysethesia
Description: as for outcome 5
Time Frame: Baseline, Week 2 and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Unit on a scale
  Baseline (n = 44, 46, 45) | 5.7 (2.02) | 6.1 (2.35) | 6.6 (1.96)
  Week 2 (n = 42, 41, 43) | 4.8 (2.45) | 5.3 (2.83) | 5.9 (2.40)
  Week 4 (n = 42, 38, 42) | 4.9 (2.34) | 5.4 (2.84) | 5.9 (2.63)
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -0.35, 90% CI 2-sided [-1.09 to 0.39], Standard Error of Mean 0.45
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -0.24, 90% CI 2-sided [-1.00 to 0.51], Standard Error of Mean 0.45

9. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) - Total Score
Description: as for outcome 5
Time Frame: Baseline, Week 2 and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Unit on a scale
  Baseline (n = 44, 45, 45） | 40.6 (17.33) | 53.4 (19.35) | 50.7 (16.87)
  Week 2 (n = 42, 40, 34) | 34.2 (17.39) | 44.6 (24.64) | 44.7 (18.11)
  Week 4 (n = 42, 37, 42) | 34.7 (19.40) | 42.7 (27.23) | 44.5 (20.18)
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -0.27, 90% CI 2-sided [-5.12 to 4.57], Standard Error of Mean 2.92
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -5.61, 90% CI 2-sided [-10.57 to -0.66], Standard Error of Mean 2.99

10. Secondary Outcome: Patient's Global Impression of Change Score (PGIC).
Description: Participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse) at week 4. The PGIC was combined to produce a 3-point scale, "Improved", "No Change" and "Worse".
Time Frame: Baseline, Week 2, and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Number of participants
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Number of participants
  Improved (Baseline, n = 43, 46, 45) | 20 | 11 | 16
  Improved (Week 2, n = 42, 41, 43) | 27 | 30 | 26
  Improved (Week 4, n = 42, 38, 42) | 28 | 27 | 24
  No change (Baseline, n = 43, 46, 45) | 19 | 30 | 25
  No change (Week 2, n = 42, 41, 43) | 10 | 7 | 13
  No change (Week 4, n = 42, 38, 42) | 12 | 9 | 14
  Worse (Baseline, n = 43, 46, 35) | 4 | 5 | 4
  Worse (Week 2, n = 42, 41, 43) | 5 | 4 | 4
  Worse (Week 4, n = 42, 38, 42) | 2 | 2 | 4
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Proportional Odds Logistic Regression including all data up to week 4; Test type: Superiority or Other; Odds Ratio (OR) = 0.70, 90% CI 2-sided [0.34 to 1.45]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Proportional Odds Logistic Regression including all data up to week 4; Test type: Superiority or Other; Odds Ratio (OR) = 0.50, 90% CI 2-sided [0.24 to 1.07]

11. Secondary Outcome: Daily Sleep Interference Scale Score (DSIS).
Description: Participant rated 11-point Likert scale ranging from 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep) during past 24-hour period. Higher score indicates a greater level of sleep disturbance. Self-assessment performed daily on awakening prior to taking study medication. This score was measured as a weekly average.
Time Frame: Baseline, Week 1, Week 2, Week 3 and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: number on a scale
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
number on a scale
  Baseline (n = 44, 46, 45) | 4.7 (2.42) | 5.6 (2.38) | 4.9 (2.29)
  Week 1 (n= 44, 46, 44) | 4.1 (2.29) | 4.7 (2.55) | 4.7 (2.46)
  Week 2 (n = 43, 44, 40) | 4.0 (2.33) | 4.1 (2.74) | 4.7 (2.41)
  Week 3 (n = 38, 40, 41) | 3.6 (2.28) | 4.4 (2.71) | 4.3 (2.49)
  Week 4 (n = 41, 38, 39) | 3.4 (2.13) | 4.2 (2.82) | 4.3 (2.51)
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -0.59, 90% CI 2-sided [-1.16 to -0.02], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -1.00, 90% CI 2-sided [-1.57 to -0.43], Standard Error of Mean 0.34

12. Secondary Outcome: Total Amount of Rescue Medication Per Week
Description: Total amount of rescue medication participants take per week
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
mg
  Baseline (n = 44, 46, 45) | 2726 (4310) | 3398 (5723) | 1863 (3684)
  Week 1 (n = 44, 46, 45) | 2272 (4043) | 2897 (5605) | 1694 (3425)
  Week 2 (n = 44, 45, 44) | 1669 (3248) | 2952 (5488) | 1391 (3238)
  Week 3 (n = 42, 42, 43) | 1851 (3228) | 1885 (4918) | 1306 (3308)
  Week 4 (n = 42, 38, 43) | 1617 (2945) | 2328 (5256) | 1372 (3307)
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = 192, 90% CI 2-sided [-1161 to 1544], Standard Error of Mean 816
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Mixed Models Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = 611, 90% CI 2-sided [-735 to 1956], Standard Error of Mean 812

13. Secondary Outcome: Number of Days Participants Take Rescue Medication
Description: Number of days participants take rescue medication per week.
Time Frame: Baseline, Week 1, Week 2, Week 3 and Week 4
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
days
  Baseline (n = 44, 46, 45) | 2.8 (3.49) | 2.1 (3.02) | 1.6 (2.60)
  Week 1 (n = 44, 46, 45) | 2.3 (3.16) | 1.8 (2.74) | 1.5 (2.50)
  Week 2 (n = 44, 45, 44) | 2.0 (3.08) | 1.7 (2.63) | 1.2 (2.25)
  Week 3 (n = 42, 42, 43) | 2.1 (3.00) | 1.2 (2.35) | 1.0 (2.10)
  Week 4 (n = 42, 38, 43) | 1.9 (2.80) | 1.6 (2.55) | 1.1 (2.28)

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Withdrawals Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect.
Time Frame: Screening to Day 36, and Day 64
Population: The safety analysis set included all participants who receive at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Participants
  Participants with TEAEs | 16 | 24 | 17
  Participants with SAE | 1 | 1 | 0
  Withdrawals due to AEs | 1 | 5 | 2

15. Secondary Outcome: Number of Participants With Laboratory Test Values of Potential Clinical Importance
Description: The total number of participants with laboratory test abnormalities (without regard to baseline abnormality) was assessed. Clinical laboratory tests included hematology, chemistry, urinalysis and some other tests.
Time Frame: Screening, Day 1, Day 15 and Day 29
Population: The safety analysis set included all participants who receive at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Participants | 38 | 35 | 37

16. Secondary Outcome: Fasted Total Cholesterol Values
Description: Percentage Change from Baseline in Fasted Total Cholesterol values
Time Frame: Baseline, Week 2 and Week 4
Population: The safety analysis set included all participants who receive at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Percent change
  Week 2 (n = 41, 37, 41) | 3.46 (12.279) | -1.45 (10.242) | -0.43 (14.271)
  Week 4 (n = 40, 33, 39) | 6.59 (15.618) | -0.11 (10.023) | -1.71 (14.242)
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Mixed Model Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = 7.99, 90% CI 2-sided [2.98 to 13.01], Standard Error of Mean 3.03
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Mixed Model Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = 0.75, 90% CI 2-sided [-4.46 to 5.95], Standard Error of Mean 3.14

17. Secondary Outcome: Fasted Low Density Lipoprotein (LDL) Cholesterol
Description: Percentage Change from Baseline in LDL cholesterol Friedewald by PEG
Time Frame: Baseline, Week 2 and Week 4
Population: The safety analysis set included all participants who receive at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Perecent change
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Number analyzed (Participants) | 44 | 46 | 45
Perecent change
  Week 2 (n = 38, 34, 39) | 8.17 (23.849) | -1.73 (14.496) | 0.81 (22.900)
  Week 4 (n = 37, 31, 36) | 13.61 (29.729) | 0.85 (13.512) | 1.48 (19.804)
Statistical Analysis 1: Comparison: PF-05089771 150 mg BID vs Placebo; Statistical analysis is only for Week 4. Mixed Model Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = 11.55, 90% CI 2-sided [2.94 to 20.17], Standard Error of Mean 5.19
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis is only for Week 4. Mixed Model Repeated Measures analysis including all data up to Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = -2.42, 90% CI 2-sided [-11.38 to 6.54], Standard Error of Mean 5.40

18. Secondary Outcome: Plasma Concentration of PF-05089771
Description: All participants in this group were analysed. Only plasma PK concentration of PF-05089771 was analysed.
Time Frame: Baseline, Week 2 and Week 4
Population: The PK concentration analysis set included all randomized participants who received at least one dose of study medication and who had at least 1 measurable concentration.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PF-05089771 150 mg BID
Number analyzed (Participants) | 44
ng/ml
  Baseline (n = 43) | NA (NA) — No Mean/SD at baseline. No subject had PK concentration value above lower limit of quantification at baseline in both groups. Summary statistics are not presented.
  Week 2 (n = 41) | 7673 (4861)
  Week 4 (n = 41) | 8784 (5749)

ADVERSE EVENTS:
Time Frame: From first dose of placebo run-in until 28 days after last dose of placebo run-out, an average of 3 months.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or 1 participant may have experienced both an AE and SAE during the study. All treated participants were included in the analysis.
Arm/Group | PF-05089771 150 mg BID | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/44 | 1/46 | 0/45
Other Adverse Events (participants affected / at risk) | 3/44 | 12/46 | 10/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05089771 150 mg BID (N=44) | Pregabalin (N=46) | Placebo (N=45)
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PF-05089771 150 mg BID (N=44) | Pregabalin (N=46) | Placebo (N=45)
Nausea (Gastrointestinal disorders) | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 5 | 2
Headache (Nervous system disorders) | 2 | 3 | 4
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/17 | 1/19 | 0/14 — AE specific to female participants. Hence the number of participants at risk refers to number of female participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.